CLINICAL TRIAL: NCT00810082
Title: Randomized ActiveStep Clinical Evaluation
Acronym: RACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TDI001
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Fall Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Standard physical therapy for fall prevention
  Interventions: Other: Standard Physical Therapy for Fall Prevention
- Group B (Experimental): Physical therapy for fall prevention that includes ActiveStep
  Interventions: Device: ActiveStep; Other: Standard Physical Therapy for Fall Prevention

INTERVENTIONS:
Device: ActiveStep — ActiveStep™ is a training simulator. The system uses a computer-controlled treadmill to recreate life-like dynamic balance challenges such as slipping and tripping in a safe, controlled environment.
  Arms: Group B
Other: Standard Physical Therapy for Fall Prevention — Standard physical therapy for fall prevention

SUMMARY:
The purpose of this study is to learn if using the ActiveStep™ treadmill reduces the number and severity of falls in older adults. This is a pilot study. The information collected will be used to support a grant application for a large multi-center trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* Referred for balance training

Exclusion Criteria:

* Age < 65

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon D Lurie, MD, MS, Principal Investigator — Dartmouth College; Richard M Greenwald, PhD, Principal Investigator — Simbex Corporation
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Alice Peck Day Memorial Hospital, Lebanon, New Hampshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from two sites, each a physical therapy clinic in a hospital setting.
Groups:
- Standard Physical Therapy Only: Physical therapy for fall prevention according to the clinician's standard practice.
- Physical Therapy Incuding ActiveStep: Physical therapy for fall prevention according to the therapist's standard practice but with the addition of the ActiveStep treadmill. The ActiveStep is a treadmill incorporating a harness safety device. It is integrated with a computer controlled by the therapist that produces perturbations simulating trips and slips. The purpose is to train the patient how to respond to the perturbations without falling.
Period: Overall Study
Arm/Group | Standard Physical Therapy Only | Physical Therapy Incuding ActiveStep
Started | 34 | 31
Completed | 34 | 27
Not Completed | 0 | 4
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Physical Therapy Only | Physical Therapy Incuding ActiveStep | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.2 (7.65) | 81.1 (7.53) | 80.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 14 | 37
  Male | 11 | 17 | 28
Region of Enrollment [Number; unit: participants]
  United States | 34 | 31 | 65

OUTCOME MEASURES:

1. Primary Outcome: Participants With at Least One Fall
Description: Subjects who had at least one fall subsequent to treatment.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Standard Physical Therapy Only | Physical Therapy Incuding ActiveStep
Number analyzed (Participants) | 34 | 27
participants | 11 | 5

ADVERSE EVENTS:
Arm/Group | Standard Physical Therapy Only | Physical Therapy Incuding ActiveStep
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/31
Other Adverse Events (participants affected / at risk) | 0/34 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No